CLINICAL TRIAL: NCT06181487
Title: Effects of High-Intensity Functional Training on Physical Fitness and Jumping Difficulty Movement Among University Male Wushu Routine Athletes in China
Brief Title: Effects of High-Intensity Functional Training on Physical Fitness and Jumping Difficulty Movement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Wang Xinzhi, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Wang Xinzhi
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Athletes
Keywords: high intensity functional training

STUDY DESIGN:
Who Masked: Participant
Masking Description: In order to avoid mutual interference between the experimental group and the control group, a blinding method needs to be used in the study. In this study, a single blind experiment will be conducted to blind the participating athletes. During the sample grouping process, participating athletes will not know the specific grouping situation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will undergo 60 minutes of high-intensity functional training.
  Interventions: Other: High Intensity Functional Training
- Control group (No Intervention): The control group will follow the curriculum standards set by the Sports University.

INTERVENTIONS:
Other: High Intensity Functional Training — 12 weeks of high-intensity functional training, 3 times/week. Each class lasts 60 minutes, including warm-up, physical training, and cool down.
  Arms: Experimental group

SUMMARY:
While prior research indicates the efficacy of High-Intensity Functional Training (HIFT) in improving physical fitness and skill performance across various sports , its effects on Wushu routine athletes still need to be determined. This study aims to explore the impact of high-intensity functional training on the physical fitness and jumping difficulty of Wushu routine athletes, providing valuable insights for coaches and athletes to optimize training plans. Coaches or sports researchers can use this knowledge to manage the training load of athletes better, thereby helping Wushu athletes achieve better results in Wushu jumping difficulty movements training.

DETAILED DESCRIPTION:
In this study, the intervention design part of the researchers referred to Greg Glassman's (2010) "CrossFit training guide" and designed a high-intensity functional training program based on the characteristics of wushu routines . This study employs a Cluster Randomized Controlled Trial (CRCT) design. The experimental period of this study is 12 weeks, three times per week. The training lasts 1.5 hours, including one hour of physical fitness training and half an hour of specialized technical training. The sample for this study is male Wushu routine athletes from the Hebei Institute of Physical Education and Hebei Normal University, with 60 participants. Athletes were randomly assigned to two different training locations and divided into experimental and control groups. The specialized skills training content of the two groups is the same, with the only difference being the physical training part. The experimental group received high-intensity functional training, while the control group maintained routine training. In addition, the specific content of routine training for the control group is the school's standard training plan. The dependent variables to be measured in this study are physical fitness (strength, power, speed, endurance, and flexibility) and jumping difficulty movements (Flying Kick, Whirl Wind Kick, Outward Leg Swing in Flight, and Side Somersaults). This study measured the dependent variable three times throughout the intervention: baseline before the experimental intervention, post-test 1 after 6 weeks, and post-test 2 after 12 weeks. Finally, statistical analysis was conducted on the three test results.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Aged 18-23 years old.
* Health.
* No experience of high-intensity functional training.

Exclusion Criteria:

* Athletes with physical surgery.
* Have high-intensity functional training experience.

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Effects of strength among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Record the number of push-ups in 1 min.
Effects of power among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Measure the distance of the standing long jump with a measuring tape in centimeters (cm).
Effects of endurance among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Recorded the number of jumping ropes in 1 min.
Effects of speed among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Use a stopwatch to record the duration of the subject's 30 m sprint (in seconds).
Effects of flexibility among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Use the sit-and-reach box. The score is recorded as the point where their fingertips reach the measurement scale. The range of motion is measured in cm.
Effects of Flying Kick among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Record the flying kick using a high-speed camera and score it by experts.
Effects of Whirlwind Kick among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Record Whirl Wind Kick using a high-speed camera and score it by experts.
Effects of Outward Leg Swing in Flight among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Record outward leg swing in flight using a high-speed camera and score it by experts.
Effects of Side Somersaults among college students | Baseline, post-test 1 after 6 weeks and post-test 2 after 12 weeks
  Record side somersaults using a high-speed camera and have experts score them.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Geok Soh, Study Director — professor
Locations (1):
- Kim Geok Soh, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bird, S., & Barrington-Higgs, B. (2010). Exploring the Deadlift. Strength & Conditioning Journal, 32(2), 46. https://doi.org/10.1519/SSC.0b013e3181d59582
- [Background] Crossley KM, Zhang WJ, Schache AG, Bryant A, Cowan SM. Performance on the single-leg squat task indicates hip abductor muscle function. Am J Sports Med. 2011 Apr;39(4):866-73. doi: 10.1177/0363546510395456. Epub 2011 Feb 18. PMID 21335344
- [Background] Feito, Y., Brown, C., & Olmos, A. (2019). A content analysis of the High-Intensity Functional Training Literature: A look at the past and directions for the future. Human Movement, 20(2), 1-15.
- [Background] Glassman, G. (2010). The CrossFit training guide. CrossFit Journal, 30(1), 1-115
- [Result] Ambrozy T, Rydzik L, Kwiatkowski A, Spieszny M, Ambrozy D, Rejman A, Koteja A, Jaszczur-Nowicki J, Duda H, Czarny W. Effect of CrossFit Training on Physical Fitness of Kickboxers. Int J Environ Res Public Health. 2022 Apr 8;19(8):4526. doi: 10.3390/ijerph19084526. PMID 35457394